CLINICAL TRIAL: NCT01852240
Title: Periodontal Disease as a Risk Indicator for Erectile Dysfunction - A Cross-sectional Study on 100 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Kristina Bertl, DMD, MSc, Medical University of Vienna
Other Study IDs: Perio&ED
Record Dates: First submitted 2013-05-06; First posted 2013-05-13 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Erectile Dysfunction; Periodontitis; hsCRP
MeSH Terms: conditions — Erectile Dysfunction; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- erectile dysfunction: Inclusion criteria:
  * male patients with ED defined by an IIEF-5 score of ≤ 21
  * age between 18-45a
  Exclusion criteria:
  * systemic diseases (e.g. diabetes mellitus, heart disease, hypertension, neurological disorders etc.)
  * pure psychogenic (non-organic) ED with good spontaneous / nightly erections
  * periodontal treatment within the last 3 months
  * antibiotic intake within the last 3 months

SUMMARY:
Background Increased levels of C reactive protein (CRP) can be found not only within individuals with periodontal diseases and those with atherosclerotic alterations but also have been proved in men with erectile dysfunction (ED). NO seems to be the key mediator in the endothelial-derived vasodilation and penile erection.

The incidence of ED increases in patients with diabetes, hypertonia, hypercholesteremia, cardiovascular diseases and renal failure. First evidence suggests that there is a relationship between periodontal disease and ED as well. Due to slow progression of chronic periodontal disease (0.3-0.5mm attachment loss/year) it can be assumed, that periodontal disease exists mainly before ED develops.

Specific Aims This cross-sectional study aims to assess the incidence of periodontal disease in male individuals with ED. A possible correlation between severity of periodontal disease, level of systemic hs-CRP and ED will be assessed. Additionally, further risk factors for endothelial dysfunction, such lipid values, will be determined and regarded in the analysis.

Hypothesis The investigators assume, that severity of ED correlates with severity of periodontal disease as well as with systemic involvement assessed by CRP-levels. In detail, the investigators hypothesize, that severity of ED (assessed by the questionnaire "International Index of Erectile Function") correlates with the mean probing depth and the level of systemic hs-CRP.

Material and Methods

1. st appointment: In the present cross-sectional study 100 male patients with ED will be included. Patients who visit the urological department (Rudolfstiftung) for ED-treatment will be asked to participate. The erectile dysfunction will be assessed by means of a questionnaire (International Index of Erectile Function - IIEF-5). Urologic examination. The following blood parameters will be assessed: testosterone, prolactin, hs-CRP, tumor necrosis factor (TNF)-alpha, Interleukin-1, total cholesterol, LDL, HDL, HbA1c and fasting glucose.
2. nd appointment: At the department of Oral Surgery (Bernhard Gottlieb School of Dentistry) the periodontal situation and the index of decayed-missing-filled permanent teeth (DMFT) index of the patients will be determined. A panoramic radiograph for assessment of alveolar bone loss and a periodontal status (probing depth, recession, bleeding- and plaque-indices) will be performed. The observer at the dental clinic will have no information on the severity of the ED (observer blinded).

ELIGIBILITY:
Inclusion criteria:

* male patients with ED defined by an IIEF-5 score of ≤ 21
* age between 18-45a

Exclusion criteria:

* systemic diseases (e.g. diabetes mellitus, heart disease, hypertension, neurological disorders etc.)
* pure psychogenic (non-organic) ED with good spontaneous / nightly erections
* periodontal treatment within the last 3 months
* antibiotic intake within the last 3 months

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In the present cross-sectional study 100 male patients with ED will be included. Patients who visit the urological department (Rudolfstiftung) for ED-treatment will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
IIEF-questionnaire-value | 1 day (cross-sectional, patients will not be followed up)
  IIEF-questionnaire-value - indicates severity of erectile dysfunction
high sensitive C-reactive protein | 1 day (cross-sectional, patients will not be followed up)
  blood value (mg/dl), assess correlation to IIEF-value
severity of periodontal disease | 1 day (cross-sectional, patients will not be followed up)
  mean pocket depth (mm), assess correlation to IIEF-value

CONTACTS AND LOCATIONS:
Locations (1):
- Krankenanstalt Rudolfstiftung, Vienna, Austria